CLINICAL TRIAL: NCT05785234
Title: The Effects of Sufentanil-remimazolam vs. Remifentanil-remimazolam Total Intravenous Anesthesia on Postoperative Pain in Laparoscopic-assisted Gastrectomy - A Randomized, Controlled Study-
Brief Title: The Effects of Sufentanil vs. Remifentanil in Total Intravenous Anesthesia With Remimazolam on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2022-1606
Record Dates: First submitted 2023-02-28; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanil-remimazolam group (Experimental): The sufentanil-remimazolam group receives total intravenous anesthesia with sufentanil-remimazolam.
  Interventions: Drug: sufentanil-remimazolam group
- Remifentanil-remimazolam group (Active Comparator): The remifentanil-remimazolam group receives total intravenous anesthesia with remifentanil-remimazolam.
  Interventions: Drug: remifentanil-remimazolam group

INTERVENTIONS:
Drug: sufentanil-remimazolam group — Induction of general anesthesia with 6mg·kg-1·h-1 of remimazolam combined with 0.5 ng·ml-1 of sufentanil. Maintenance of general anesthesia with 1-2mg·kg-1·h-1 of remimazolam combined with 0.2 - 0.6 ng·ml-1 of sufentanil.
  Arms: Sufentanil-remimazolam group
Drug: remifentanil-remimazolam group — Induction of general anesthesia with 6mg·kg-1·h-1 of remimazolam combined with 4 ng·ml-1 of remifentanil. Maintenance of general anesthesia with 1-2mg·kg-1·h-1 of remimazolam combined with 2-6 ng·ml-1 of remifentanil.
  Arms: Remifentanil-remimazolam group

SUMMARY:
In this study, the investigators evaluate the effect of total intravenous anesthesia using sufentanil-remimazolam and remifentanil-remimazolam on postoperative pain in patients undergoing laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. 20years or older
2. Scheduled for laparoscopic-assisted gastrectomy
3. American Society of Anesthesiologists(ASA) physical status I and III

Exclusion Criteria:

1. Emergency operation
2. Patients with a history of severe hypersensitivity reaction to dextran 40
3. Patients who cannot use patient controlled analgesia(PCA)
4. Patients with morbid obesity [body mass index (BMI) >35 kg/m2]
5. Patients with history of uncontrolled hypertension (diastolic BP >110mmHg) or DM
6. Patients with history of heart failure (unstable angina, congestive heart failure)
7. Patients with history of liver failure, renal failure, allergic to medicine
8. Patients with history of cerebrovascular disease (cerebral hemorrhage, cerebral ischemia)
9. Patients with history of uncontrolled psychiatric disease (PTSD, anxiety, depression)
10. Patients with obstructive sleep apnea
11. Patients who cannot read the consent form (examples: Illiterate, foreigner)
12. Patients who withdraw the consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Total consumption of fentanyl in 24 hours after surgery | after 24 hours postoperative period
  To investigate the effect of total intravenous anesthesia with intraoperative sufentanil-remimazolam and remifentanil-remimazolam on postoperative pain, total cumulative dose of fentanyl was measured for the first postoperative 24 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Joon Bai, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea